CLINICAL TRIAL: NCT03451448
Title: Combined Magnetic Resonance Coronary Angiography and Positron Emission Tomography in Patients With Coronary Artery Disease
Brief Title: PET MRI in Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 17/SS/0151
Record Dates: First submitted 2018-02-23; First posted 2018-03-01 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Coronary Artery Disease
Keywords: PET/MRI; ultra-small-superparamagnetic particles
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy volunteers: Healthy volunteers to undergo MRI using USPIO contrast
  Interventions: Diagnostic Test: MRI
- Stable coronary artery disease: Patients with coronary artery disease without recent (3 months) acute coronary syndrome or revascularisation
  Interventions: Diagnostic Test: PET/MRI
- Recent acute coronary syndrome: Patients with recent (3 months) type 1 myocardial infarction
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — PET/MRI with USPIO contrast
  Groups: Recent acute coronary syndrome; Stable coronary artery disease
Diagnostic Test: MRI — MRI with USPIO contrast
  Groups: Healthy volunteers

SUMMARY:
This study will assess the use of position emission tomography/magnetic resonance imaging (PET/MRI) using ultra-small-superparamagnetic particles of iron oxide (USPIO) as a contrast agent in patients with coronary artery disease.

DETAILED DESCRIPTION:
Positron emission tomography/magnetic resonance imaging (PET/MRI) has the potential to provide detailed information on coronary artery anatomy, the presence of coronary artery stenosis, the composition of atherosclerotic plaque using MRI tissue characterisation and information about the underlying biological processes using targeted PET tracers. Ultra-small-superparamagnetic particles of iron oxide (USPIO) have a long blood pool half-life so are an ideal contrast agent for PET/MRI imaging.

This study will assess the use of PET/MRI with USPIO in patients with stable coronary artery disease and recent acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers to undergo MRI imaging will be over the age of 18 years and able to provide informed consent.
* Patients with coronary artery disease to undergo PET/MRI will have multi-vessel disease (≥2 vessel coronary artery disease with ≥ 50% cross-sectional luminal stenosis).
* able to provide informed consent
* over the age of 40 years

Exclusion Criteria:

* inability or unwillingness to undergo magnetic resonance imaging or positron emission tomography
* renal failure (Serum creatinine >200 umol/L or estimated glomerular filtration rate <30 mL/min
* hepatic failure
* pregnancy
* inability to provide informed consent
* contraindications to undergoing MRI scanning
* contraindications to contrast agents not included above including evidence of iron overload, known allergy to constituents of the contrast agents, and anaemia not caused by iron deficiency

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers to undergo MRI.
  Patients with stable coronary artery disease or recent acute myocardial infarction to undergo PET/MRI
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
PET/MRI findings | Immediately after PET/MRI scan
  The primary endpoint will be the difference in MRI and PET characteristics of atherosclerotic plaques in patients with and without recent acute coronary syndromes.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Williams, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided